CLINICAL TRIAL: NCT04191642
Title: Correlation of NLRP3 With Cognitive Dysfunction Early After Heart Valve
Brief Title: Correlation of NLRP3 With Cognitive Dysfunction Early After Heart Valve Replacement Surgery
Status: Completed | Type: Observational
Sponsor: General Hospital of Ningxia Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: Magang2018-020
Record Dates: First submitted 2019-11-27; First posted 2019-12-10 (Actual); Last update posted 2021-09-01 (Actual); Status verified 2021-08

CONDITIONS: Inflammasomes; Cognitive Dysfunction; Pyrin Domain-Containing 3 Protein; Postoperative Complications
Keywords: Inflammasomes; Interleukin-18; Interleukin-1; NLR Family, Pyrin Domain-Containing 3 Protein; Postoperative cognitive dysfunction
MeSH Terms: conditions — Cognitive Dysfunction; Postoperative Complications; Postoperative Cognitive Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Before induction of anesthesia, at the end of the operation, 7 days after the operation, peripheral venous blood was sampled to measure IL-1B, IL-18 and NLRP3 inflammatory protein expression in peripheral blood monocytes.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The investigators decided to assess the prognostic value of NLRP3 inﬂammasome level in early after heart valve replacement surgery and whether it was related to postoperative cognitive dysfunction. Study population included 90 subjects. Neuropsychological tests were administrated one day before surgery and seven days after surgery. Before induction of anesthesia, before the end of the operation, 7 days after the operation, peripheral venous blood was sampled to measure IL-1B, IL-18 and NLRP3 inflammatory protein expression in peripheral blood monocytes. Analyze the data and draw conclusions.

DETAILED DESCRIPTION:
90 consecutive patients scheduled for mitral valve replacement or aortic valve replacement under moderate hypothermic CPB gave written informed consent and were enrolled in this study.

In the operating room, patients received routine monitoring. Systemic arterial blood pressure was measured via radial artery catheterization. After induction of anesthesia, a central venous catheter was inserted for monitoring central venous pressure (CVP) and fluid management. Baseline readings of hemodynamics were taken every 5 to 10 min after radial artery cannulation was completed.

Induction of anesthesia was performed with target-controlled infusion of propofol. All patients received an infused scheme of several steps that started from a target plasma concentration (Cp) of 0.5 mg/mL that was increased stepwise by 0.5 mg/mL until the patient fell asleep and maintain BIS at 40-60. The interval between each step was 3 min. After loss of consciousness, cisatracurium (0.2 mg/kg) and fentanyl (10-15 mg/kg) were infused in all groups. The trachea was intubated and the lungs were ventilated with oxygenenriched air (fraction of inspired oxygen 0.6) to an end-tidal carbon dioxide partial pressure of 35 to 45 mmHg. The propofol target Cp was adjusted according to BIS. Intermittent IV boluses of fentanyl (10-15 mg/kg) were administered according to blood pressure and heart rate (HR) at the following time points: before the skin incision, before the onset of CPB, and after separation from CPB, for a total dose of 40 to 50 mg/kg. All patients received infusion of cisatracurium at 0.1 mg/kg/h throughout the surgery.

Surgery was conducted on all patients via a standard median sternotomy approach. Porcine heparin was administered at a dose of 300 IU/kg and supplemented when required to maintain an activated coagulation time of at least 480 s during CPB. Heparin was neutralized with 1 mg of protamine/100 IU of heparin administered after separation from CPB. Body temperature was cooled to 30℃-32℃ on CPB (moderate hypothermia). All patients were treated with an intermittent antegrade infusion of cooled high-potassium blood cardioplegia during continuous aortic cross-clamping (ACC) using a nonpulsatile flow rate of 1.8 to 2.8 L/min/m2 and a membrane oxygenator to keep the mixed venous saturation at more than 75% during CPB. Phenylephrine (bolus, 20-100 mg) or epinephrine (0.1 mg/kg/min) or both were used to restore systemic vascular resistance, and MAP was maintained at a target range of 60 to 80 mmHg. Patients were warmed to a bladder temperature of 36.5℃ before separation from CPB, with the highest temperature not exceeding 37℃. Blood remaining in the CPB circuit and from the surgical field was collected in a cell-saving device. After centrifuging and washing, it was infused to the patient within 4 hours after CPB. Hematocrit was maintained at more than 25%, with the addition of blood as necessary. Insulin therapy was initiated during the surgery to treat serum blood glucose levels higher than 150 mg/dL. Hemodynamic (pre- or post-CPB) management aimed to keep MAP at 60 to 100 mmHg. Hypertension was treated with an additional bolus dose of fentanyl (0.2-0.3 mg) or with nitroglycerin (0.1-0.5 mg/kg/min or with both). Hypotension was treated with fluid intake (including crystalloids, colloids, and blood products) or vasoactive drug administration (phenylephrine IV, 20-100 mg or concomitant use of epinephrine, o 0.1 mg/min). The vasoactive drug dosage, fluid intake, and output (urine and blood loss) were recorded when the surgery was finished.

As the surgeons began to close the skin, a 0.08 mg/kg bolus dose of midazolam was given intravenously and the infusion of propofol was stopped. After the surgery, all patients were admitted to the surgical intensive care unit (ICU). The patients were extubated when they were able to sustain adequate spontaneous respiration and required minimal oxygen support, as reflected by normal arterial blood gas levels. The patients then were discharged from the ICU when they were hemodynamically stable with blood gas variables within the normal range and when they did not need inotropic or oxygen support. The tracheal extubation time and the length of the ICU stay were recorded. For all patients, hemodynamic measurements were made and recorded at the following times: Before induction of anesthesia, before skin incision, after sternotomy, at the cessation of CPB (CPB-cessation), and at 1 (Post-CPB 1 h), 2 (Post-CPB 2 h), and 4 (Post-CPB 4 h) hours after CPB. At pre-incision, CPB-cessation, Post-CPB 2 h, and PostCPB 4 h, the radial arterial blood was sampled for blood gas analysis, as well as blood glucose and lactic acid analyses. Before induction of anesthesia, at the end of the operation, 7 days after the operation, peripheral venous blood was sampled to measure IL-1B, IL-18 and NLRP3 inflammatory protein expression in peripheral blood monocytes.

Neuropsychological tests were administrated one day before surgery and seven days after surgery for all patients in a quiet place of the general wards. Neuropsychological tests included seven tests with nine subscales. Specific tests used were as follows: MMSE, Trail Making (A/B), Stroop Color- Word, Rey Auditory Verbal Learning Test, WAIS Digit Symbol Substitution Test, WAIS Digit Span, Verbal fluency test. Two psychologists carried out these tests. During the study phase, testing was performed and scored in a standardized manner in order to minimize inter-examiner difference. Repeat assessments for each patient were conducted by the same examiner. Parallel forms of tests were used in a randomized manner in sequential testing in order to minimize practice effect. Performance on each test was compared with cognitive test data of control subjects. A low test score was defined when the score was ≥ 2 SD lower than control subjects. For tests in which a higher score indicates decrement in performance, a score ≥ 2 SD higher than control subjects was considered as "low test score." Patients were defined as having preoperative cognitive impairment if they had low test scores on two or more tests.

For patients, preoperative scores were compared with postoperative test results, subtracted the average practice effect from these changes, and then divided the result by the control-subject SD to obtain a Z score for each test. The test results were adjusted so that a positive Z score indicated deterioration from the baseline test. The Z scores of all tests in an individual patient were then summarized and divided by the SD for this sum of Z scores in the control subjects, creating a combined Z score. A patient was defined as having POCD when two Z scores in individual tests or the combined Z score were 1.96 or more.

Statistical analysis A continuous outcome was expressed as the mean ± SE, while a categorical outcome was expressed as percentages or frequencies. Differences in continuous and categorical outcomes were tested using the one-way analysis of variance and Chi square analysis, respectively. The unpaired Student t test, paired T test, analysis of variance and Pearson correlation analysis were performed on normally distributed data. Case-control differences in nominal data were evaluated with the Chi square test. Multivariate Cox regression analysis was done for predictors of adverse events. The NLRP3 level, IL-1B, IL-18 and neurobehavioral scores were compared using ROC curves. Kaplan-Meier curves were used for correlation with POCD. All statistical analyses were performed with SPSS 21.0 (IBM Inc.) and P < 0.05 was considered signifcant.

ELIGIBILITY:
Inclusion Criteria:

* Patients were included if they had an American Society of Anesthesiologists status of II or III and older than 60 years old.

Exclusion Criteria:

* A preoperative history of liver or kidney dysfunction, peripheral vascular disease, diabetes mellitus, or arterial hypertension;
* Ischemic cerebrovascular disease;
* A history of an acute or evolving myocardial infarction or presentation with a left ventricular ejection fraction (LVEF) of less than 45%;
* Obesity (body mass index 430 kg/m2);
* Moderate or severe atherosclerotic lesions in the ascending aorta or carotid artery stenosis confirmed by preoperative ultrasonography
* Patients requiring re-exploration after surgery or a total CPB time more than 115 min
* Patients requiring highdose pharmacologic support (phenylephrine 4 100 mg bolus, or epinephrine 4 0.1mg/kg/min or both) to maintain hemodynamic stability (mean arterial pressure [MAP] more than 60 mmHg)

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Elderly heart surgery patients
Sampling Method: Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2021-01-30 (Actual); Study Completion 2021-01-30 (Actual)

PRIMARY OUTCOMES:
The correlation between peripheral blood NLRP3 inﬂammasome level and incidence of postoperative cognitive dysfunction | The day before surgery, 7 days after surgery
  Peripheral venous blood was sampled to measure NLRP3 inﬂammasome expression.
  POCD was defined by Z scores that based on the neuropsychological tests, and then, get the incidence of POCD.
  The method of Z scores is as follows: A patient was defined as having POCD when two Z scores in individual tests or the combined Z score were 1.96 or more.
  Neuropsychological tests included MMSE(screening method); Trail Making (A/B); Stroop Color-Word; Rey Auditory Verbal Learning Test; WAIS Digit Symbol Substitution Test; WAIS Digit Span; Verbal fluency test.
  Preoperative scores were compared with postoperative test results, subtracted the average practice effect from these changes, and then divided the result by the control-subject SD to obtain a Z score for each test. The Z scores of all tests in an individual patient were then summarized and divided by the SD for this sum of Z scores in the control subjects, creating a combined Z score.

SECONDARY OUTCOMES:
The correlation between peripheral blood IL-1B levels and incidence of postoperative cognitive dysfunction | At the end of the surgery, 7 days after surgery
  Peripheral venous blood was sampled to measure IL-1B expression.
  POCD was defined by Z scores that based on the neuropsychological tests, and then, get the incidence of POCD.
  The method of Z scores is as follows: A patient was defined as having POCD when two Z scores in individual tests or the combined Z score were 1.96 or more.
  Neuropsychological tests included MMSE(screening method); Trail Making (A/B); Stroop Color-Word; Rey Auditory Verbal Learning Test; WAIS Digit Symbol Substitution Test; WAIS Digit Span; Verbal fluency test.
  Preoperative scores were compared with postoperative test results, subtracted the average practice effect from these changes, and then divided the result by the control-subject SD to obtain a Z score for each test. The Z scores of all tests in an individual patient were then summarized and divided by the SD for this sum of Z scores in the control subjects, creating a combined Z score.
The correlation between peripheral blood IL-18 levels and incidence of postoperative | At the end of the surgery, 7 days after surgery
  Peripheral venous blood was sampled to measure IL-18 expression.
  POCD was defined by Z scores that based on the neuropsychological tests, and then, get the incidence of POCD.
  The method of Z scores is as follows: A patient was defined as having POCD when two Z scores in individual tests or the combined Z score were 1.96 or more.
  Neuropsychological tests included MMSE(screening method); Trail Making (A/B); Stroop Color-Word; Rey Auditory Verbal Learning Test; WAIS Digit Symbol Substitution Test; WAIS Digit Span; Verbal fluency test.
  Preoperative scores were compared with postoperative test results, subtracted the average practice effect from these changes, and then divided the result by the control-subject SD to obtain a Z score for each test. The Z scores of all tests in an individual patient were then summarized and divided by the SD for this sum of Z scores in the control subjects, creating a combined Z score.

CONTACTS AND LOCATIONS:
Overall Officials: Gang Ma, doctor, Study Director — Department of Anesthesiology General Hospital of Ningxia Medical University
Locations (1):
- Department of Anesthesiology, General Hospital of Ningxia Medical University, Yinchuan, Ningxia, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Afrasyab A, Qu P, Zhao Y, Peng K, Wang H, Lou D, Niu N, Yuan D. Correlation of NLRP3 with severity and prognosis of coronary atherosclerosis in acute coronary syndrome patients. Heart Vessels. 2016 Aug;31(8):1218-29. doi: 10.1007/s00380-015-0723-8. Epub 2015 Aug 20. PMID 26290166
- [Result] Meital LT, Coward AS, Windsor MT, Bailey TG, Kuballa A, Russell FD. A simple and effective method for the isolation and culture of human monocytes from small volumes of peripheral blood. J Immunol Methods. 2019 Sep;472:75-78. doi: 10.1016/j.jim.2019.04.005. Epub 2019 Jun 20. PMID 31229469
- [Result] Lenart N, Brough D, Denes A. Inflammasomes link vascular disease with neuroinflammation and brain disorders. J Cereb Blood Flow Metab. 2016 Oct;36(10):1668-1685. doi: 10.1177/0271678X16662043. Epub 2016 Aug 2. PMID 27486046
- [Result] Feinkohl I, Winterer G, Spies CD, Pischon T. Cognitive Reserve and the Risk of Postoperative Cognitive Dysfunction. Dtsch Arztebl Int. 2017 Feb 17;114(7):110-117. doi: 10.3238/arztebl.2017.0110. PMID 28302254
- [Result] Cao XZ, Ma H, Wang JK, Liu F, Wu BY, Tian AY, Wang LL, Tan WF. Postoperative cognitive deficits and neuroinflammation in the hippocampus triggered by surgical trauma are exacerbated in aged rats. Prog Neuropsychopharmacol Biol Psychiatry. 2010 Dec 1;34(8):1426-32. doi: 10.1016/j.pnpbp.2010.07.027. Epub 2010 Aug 4. PMID 20691747
- [Result] Cibelli M, Fidalgo AR, Terrando N, Ma D, Monaco C, Feldmann M, Takata M, Lever IJ, Nanchahal J, Fanselow MS, Maze M. Role of interleukin-1beta in postoperative cognitive dysfunction. Ann Neurol. 2010 Sep;68(3):360-8. doi: 10.1002/ana.22082. PMID 20818791
- [Result] Song L, Pei L, Yao S, Wu Y, Shang Y. NLRP3 Inflammasome in Neurological Diseases, from Functions to Therapies. Front Cell Neurosci. 2017 Mar 9;11:63. doi: 10.3389/fncel.2017.00063. eCollection 2017. PMID 28337127
- [Result] Murkin JM, Newman SP, Stump DA, Blumenthal JA. Statement of consensus on assessment of neurobehavioral outcomes after cardiac surgery. Ann Thorac Surg. 1995 May;59(5):1289-95. doi: 10.1016/0003-4975(95)00106-u. No abstract available. PMID 7733754
- [Result] Rudolph JL, Schreiber KA, Culley DJ, McGlinchey RE, Crosby G, Levitsky S, Marcantonio ER. Measurement of post-operative cognitive dysfunction after cardiac surgery: a systematic review. Acta Anaesthesiol Scand. 2010 Jul;54(6):663-77. doi: 10.1111/j.1399-6576.2010.02236.x. Epub 2010 Apr 15. PMID 20397979
- [Derived] Ma G, Sun P, Chen Y, Jiang X, Zhang C, Qu B, Meng X. NLRP3 inflammasome activation contributes to the cognitive decline after cardiac surgery. Front Surg. 2022 Nov 2;9:992769. doi: 10.3389/fsurg.2022.992769. eCollection 2022. PMID 36406365